CLINICAL TRIAL: NCT02891850
Title: A Prospective, Randomized, International, Multicenter, Double-arm, Controlled, Open-label Study of Riociguat in Patients With Pulmonary Arterial Hypertension (PAH) Who Are on a Stable Dose of Phosphodiesterase-5 Inhibitors (PDE-5i) With or Without Endothelin Receptor Antagonist (ERA), But Not at Treatment Goal
Brief Title: Riociguat rEplacing PDE-5i Therapy evaLuated Against Continued PDE-5i thErapy
Acronym: REPLACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18588; 2016-001067-36 (EudraCT Number)
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — riociguat; Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Riociguat (Experimental): PDE5i treatment will be stopped and riociguat treatment initiated following a defined washout period with a starting dose of 1 mg riociguat TID followed by an 8 weeks dose adjustment phase according to the approved riociguat dose adjustment scheme.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- PDE-5i (Active Comparator): Patients will continue to receive PDE5i treatment as well as other standard of care treatments at the discretion of the investigator up to Week 24. Patients in the experimental and active comparator treatment arms follow the same visit schedule.
  Interventions: Drug: Sildenafil; Drug: Tadalafil

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Film-coated tablets will be used in this study at a dosage of 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg and 2.5 mg. Tablets will be administered orally.The starting dose is 1 mg TID; the intervals between drug intakes should be 6 to 8 hours. The dosage should be increased by 0.5 mg increments in 2 week intervals to 1.5 mg, 2.0 mg, and 2.5 mg TID (maximal total daily dose).
  Arms: Riociguat
Drug: Sildenafil — Patients randomized to the control arm will continue to receive stable doses of tadalafil (daily dose 20 to 40 mg) or sildenafil (daily dose at least 60 mg) as well as other supportive treatments at the discretion of the investigator.
  Arms: PDE-5i
Drug: Tadalafil — Patients randomized to the control arm will continue to receive stable doses of tadalafil (daily dose 20 to 40 mg) or sildenafil (daily dose at least 60 mg) as well as other supportive treatments at the discretion of the investigator.
  Arms: PDE-5i

SUMMARY:
To demonstrate the effectiveness of riociguat as replacement of phosphodiesterase-5 inhibitors (PDE-5i) therapy in pulmonary arterial hypertension (PAH) patients

DETAILED DESCRIPTION:
Data from a previous single arm study (RESPITE) indicate that transition from PDE5i to riociguat may be feasible, safe and beneficial in patients not adequately responding to PDE5i.

REPLACE is a randomized controlled study to confirm the potential clinical benefit of transition from PDE5i to riociguat. Satisfactory clinical response in patients who are on a stable dose of phosphodiesterase-5inhibitors (PDE-5i) with or without endothelin receptor antagonist (ERA), but not at treatment goal will be compared between one group of patients randomized to maintain current treatment and another group where the PDE5i is replaced by riociguat.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 75 years.
* Patients with symptomatic PAH with a pulmonary vascular resistance (PVR) > 400 dyn*sec*cm-5, mean pulmonary artery pressure ≥ 25 mmHg, and pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg as assessed by the most recent right heart catheterization (RHC) from medical history prior to screening to confirm the diagnosis. Alternatively, PCWP can be replaced by left ventricular end-diastolic pressure (≤ 15 mmHg). PAH of the following types:

  * Idiopathic
  * Hereditary
  * Drug and toxin induced PAH
  * Associated with PAH due to:

    * Connective tissue disease (CTD)
    * Congenital heart disease, but only if the patient underwent surgical repair more than one year before enrolment
    * Portal hypertension with liver cirrhosis (Note: patients with clinical relevant hepatic dysfunction are excluded; see exclusions related to disorders in organ function)
* Patients who are on stable doses of a PDE-5i and ERA combination therapy or on stable PDE-5i monotherapy 6 weeks prior to and at randomization but not at treatment goal (tadalafil 20 to 40 mg once daily or sildenafil at least 60 mg daily dose).
* WHO FC III at screening and at randomization.
* 6MWD test between 165 m and 440 m at screening and at randomization.
* Stable dose of diuretics, if used, for at least 30 days prior to and at randomization.
* Patients who are able to understand and follow instructions and who are able to participate in the study for the entire study.
* Women of childbearing potential must agree to use adequate contraception when sexually active. Adequate contraception is defined as any combination of at least 2 effective methods of birth control, of which at least 1 is a physical barrier (e.g. condom with hormonal contraception like implants or combined oral contraceptives, condom with intrauterine devices). This applies beginning with signing of the informed consent form until 30 (+5) days after the last administration of study drug.
* Patients must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures.

Exclusion Criteria:

* Participation in another interventional clinical study within 30 days prior to screening.
* All types of PH (including PH-IIP) except subtypes of Dana Point Group I specified in the inclusion criteria.
* Previous treatment with riociguat.
* Pregnant women (i.e., positive serum ß-human-chorionic-gonadotropin test or other signs of pregnancy), or breast feeding women, or women with childbearing potential not using a combination of 2 effective contraception methods (as laid out in inclusion criterion) throughout the study.
* Patients with a medical disorder, condition, or history of such that would impair the patient's ability to participate or complete this study, in the opinion of the investigator.
* Relevant obstructive and restrictive or other lung diseases.
* Patients with underlying medical disorders with an anticipated life expectancy below 2 years (e.g., active cancer disease with localized and/or metastasized tumor mass).
* Cardiovascular exclusion criteria like left ventricular disease, coronary heart disease or stroke within previous 3 months.
* Patients with hypersensitivity to the investigational drug or any of the excipients.
* Patients unable to perform a valid 6MWD test (e.g., orthopedic disease, peripheral artery occlusive disease, which affects the patient's ability to walk). Note: Patients, who require walking aids, may be included if in the opinion of the investigator the walking distance is not impaired. Patients with a variance of more than 15% between the screening and the randomization (i.e., baseline) 6MWD test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (70):
- United States (17):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Sacramento, California
  - Orlando, Florida
  - Weston, Florida
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Detroit, Michigan
  - Troy, Michigan
  - Newark, New Jersey
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - Cleveland, Ohio
  - Nashville, Tennessee
  - Dallas, Texas
  - Richmond, Virginia
- Graz, Austria
- Leuven, Belgium
- Brazil (4):
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Blumenal, Santa Catarina
  - São Paulo
- Montreal, Quebec, Canada
- Prague, Czechia
- Aarhus N, Denmark
- France (2):
  - Le Kremlin-Bicêtre
  - Rouen
- Germany (12):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Würzburg, Bavaria
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Lübeck, Schleswig-Holstein
  - Berlin
  - Giessen
  - Hamburg
- Greece (2):
  - Chaïdári
  - Thessaloniki
- Italy (4):
  - Napoli, Campania
  - Rome, Lazio
  - Pavia, Lombardy
  - Palermo, Sicily
- Japan (3):
  - Nagoya, Aichi-ken
  - Sendai, Miyagi
  - Bunkyo-ku, Tokyo
- Mexico (2):
  - Culiacán, Sinaloa
  - Mexico City
- Netherlands (2):
  - Amsterdam
  - Nijmegen
- Wroclaw, Poland
- Portugal (3):
  - Almada, Lisbon District
  - Coimbra
  - Lisbon
- Seoul, South Korea
- Spain (3):
  - Las Palmas de Gran Canaria, Las Palmas
  - Barcelona
  - Toledo
- Taiwan (3):
  - Kaoshiung
  - Tainan
  - Taipei
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Clydebank, West Dunbartonshire
  - London
  - Sheffield

REFERENCES:
- [Derived] Hoeper MM, Al-Hiti H, Benza RL, Chang SA, Corris PA, Gibbs JSR, Grunig E, Jansa P, Klinger JR, Langleben D, McLaughlin VV, Meyer GMB, Ota-Arakaki J, Peacock AJ, Pulido T, Rosenkranz S, Vizza CD, Vonk-Noordegraaf A, White RJ, Chang M, Kleinjung F, Meier C, Paraschin K, Ghofrani HA, Simonneau G; REPLACE investigators. Switching to riociguat versus maintenance therapy with phosphodiesterase-5 inhibitors in patients with pulmonary arterial hypertension (REPLACE): a multicentre, open-label, randomised controlled trial. Lancet Respir Med. 2021 Jun;9(6):573-584. doi: 10.1016/S2213-2600(20)30532-4. Epub 2021 Mar 24. PMID 33773120
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 21 countries between 11-JAN-2017 (first participant first visit) and 03-MAR-2020 (last participant last visit).
Pre-assignment Details: 293 participants were screened in this study. Of these, 67 participants did not enter the treatment period (60 screening failures; 2 withdraw during screening; 2 withdraw following physician decision; 3 withdraw due to other reasons). 226 participants were randomized, of which 1 participant withdraw before treated.
Groups:
- Riociguat: Participants received BAY63-2521 tablets at a dosage of 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg, and 2.5 mg three times a day (TID) for 24 weeks, started with 1.0 mg TID, followed by a dose adjustment period of 8 weeks, then stayed at the optimal dose period of 16 weeks.
- PDE-5i: Participants remained on their current pulmonary arterial hypertension (PAH) treatment on tadalafil (20 to 40 mg/day) or sildenafil (at least 60 mg/day) for 24 weeks at the discretion of the investigator.
Period: Overall Study
Arm/Group | Riociguat | PDE-5i
Started (Treated) | 111 | 114
Completed | 104 | 107
Not Completed | 7 | 7
Not completed — Adverse Event | 3 | 0
Not completed — Death | 0 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat | PDE-5i | Total
Number analyzed (Participants) | 111 | 114 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (16.16) | 49.2 (15.64) | 49.3 (15.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 95 | 177
  Male | 29 | 19 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 31 | 63
  Not Hispanic or Latino | 75 | 80 | 155
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 17 | 19 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 86 | 89 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Satisfactory Clinical Response at Week 24
Description: The treatment is assessed as efficient (participants with satisfactory clinical response) in case at least 2 out of the following 3 criteria were fulfilled
  * 6 Minute Walking Distance increase by ≥ 10% or ≥ 30 m from baseline to Week 24
  * World Health Organization Functional Class (WHO FC) I or II at Week 24
  * N-terminal pro-brain natriuretic peptide (NT-proBNP) reduction ≥ 30% from baseline to Week 24 (NT-proBNP ratio Week 24/baseline ≤ 0.7) and in absence of the defined criteria of clinical worsening
Time Frame: At Week 24
Population: Full Analysis Set (FAS) with evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | PDE-5i
Number analyzed (Participants) | 111 | 113
Participants
  With satisfactory clinical response | 45 | 23
  Without satisfactory clinical response | 66 | 90
Statistical Analysis 1: Comparison: Riociguat vs PDE-5i; Test type: Equivalence — The hypothesis was that there was no difference in the satisfactory clinical response rates in terms of odds ratio (OR) when treated with riociguat compared with participants who remained on their previous therapy; p = 0.0007, Mantel Haenszel; Stratified by PAH category at baseline; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.526 to 5.060]

2. Secondary Outcome: Change in 6 Minute Walking Distance (6MWD) With Last Observation Carried Forward From Baseline to 24 Weeks
Description: Six-minute walk distance (6MWD) was conducted to test the physical limitations of the participant by assessing the participant's exercise capacity. The distance walked by the participant in 6 minutes was measured.
Time Frame: From baseline and up to 24 weeks
Population: Full Analysis Set (FAS) with evaluable participants
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Riociguat | PDE-5i
Number analyzed (Participants) | 111 | 113
meters (m) | 36.448 (65.9748) | 13.884 (67.1552)
Statistical Analysis 1: Comparison: Riociguat vs PDE-5i; Test type: Equivalence — The hypothesis was that there was no difference in the change of 6MWD in terms of mean difference when treated with riociguat compared with participants who remained on their previous therapy; p = 0.0542, t-test, 2 sided; Stratified by PAH category at baseline; Mean Difference (Final Values) = 22.56, 95% CI 2-sided [5.03 to 40.10]

3. Secondary Outcome: Change in N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) With Last Observation Carried Forward at Week 24
Description: N-terminal pro-brain natriuretic peptide (NT-proBNP) levels in the blood are used for screening, diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: From baseline and up to 24 weeks
Population: Full Analysis Set (FAS) with evaluable participants
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Riociguat | PDE-5i
Number analyzed (Participants) | 108 | 113
picograms per milliliter (pg/mL) | -88.234 (533.9179) | 81.414 (1267.6142)
Statistical Analysis 1: Comparison: Riociguat vs PDE-5i; Test type: Equivalence — The hypothesis was that there was no difference in the change of NT-proBNP in terms of mean difference when treated with riociguat compared with participants who remained on their previous therapy; p = 0.1067, t-test, 2 sided; Stratified by PAH category at baseline; Mean Difference (Final Values) = -169.65, 95% CI 2-sided [-426.18 to 86.88]

4. Secondary Outcome: Change in World Health Organization Functional Class (WHO FC) With Last Observation Carried Forward From Baseline to Week 24
Description: The participant's functional class was determined by using the WHO classification. Possible classes range from I (patients with pulmonary hypertension (PH) but without resulting limitation of physical activity) to IV (patients with PH with inability to carry out any physical activity without symptoms).
Time Frame: From baseline and up to 24 weeks
Population: Full Analysis Set (FAS) with evaluable participants
Measure: Mean (Standard Deviation); unit: class
Arm/Group | Riociguat | PDE-5i
Number analyzed (Participants) | 111 | 113
class | -0.5 (0.58) | -0.2 (0.62)
Statistical Analysis 1: Comparison: Riociguat vs PDE-5i; Test type: Equivalence — The hypothesis was that there was no difference in the change from baseline in WHO FC in terms of mean difference when treated with riociguat compared with participants who remained on their previous therapy; p = 0.0007, t-test, 2 sided; Stratified by PAH category at baseline; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.42 to -0.11]

5. Secondary Outcome: Number of Participants With Adjudicated Clinical Worsening at Week 24
Description: Clinical worsening was defined as death of any cause, hospitalization due to worsening pulmonary arterial hypertension (PAH) (adjudicated) or disease progression (adjudicated).
Time Frame: Up to 24 weeks
Population: Full Analysis Set (FAS) with evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | PDE-5i
Number analyzed (Participants) | 111 | 113
Participants | 1 | 10
Statistical Analysis 1: Comparison: Riociguat vs PDE-5i; Test type: Equivalence — The hypothesis was that there was no difference in the clinical worsening rates in terms of odds ratio (OR) when treated with riociguat compared with participants who remained on their previous therapy; p = 0.0047, Mantel Haenszel; Stratified by PAH category at baseline; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.013 to 0.725]

ADVERSE EVENTS:
Time Frame: The adverse events were considered to be treatment emergent if they had started or worsened after the first treatment administration and up to 2 days after end of treatment. Since maximum study duration was 24 weeks, this could be up to 24 weeks + 2 days.
Arm/Group | Riociguat | PDE-5i
All-Cause Mortality (participants affected / at risk) | 0/111 | 4/114
Serious Adverse Events (participants affected / at risk) | 8/111 | 19/114
Other Adverse Events (participants affected / at risk) | 77/111 | 72/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=111) | PDE-5i (N=114)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary arterial pressure increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Drug therapy enhancement (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=111) | PDE-5i (N=114)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (4) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal disorder (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (10) | 1 (1)
Gingival hypertrophy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 5 (8) | 5 (5)
Drug ineffective (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (7) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 2 (2)
Oedema mucosal (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobiasis (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 5 (5)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 4 (4)
Sinusitis (Infections and infestations) | 2 (2) | 6 (8)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (8)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 14 (16) | 8 (8)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (3)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 13 (19) | 6 (11)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein distension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT02891850/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT02891850/SAP_001.pdf